CLINICAL TRIAL: NCT03913403
Title: Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis: Study of Treatment's Echocardiographic Mechanisms (CLOVERS-STEM)
Brief Title: Study of Treatment's Echocardiographic Mechanisms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Montefiore Medical Center (Other); Oregon Health and Science University (Other); Vanderbilt University Medical Center (Other); Wake Forest University Health Sciences (Other); Harborview Injury Prevention and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1051075
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Sepsis
Keywords: Fluid Management; Sepsis-Induced Hypotension; Vasopressors; Cardiac Contractility
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Participants will receive 2 ECHO's and 2 Blood Draws
  Interventions: Procedure: ECHO; Procedure: Blood Draw

INTERVENTIONS:
Procedure: ECHO — Echocardiogram at baseline and 24 hours later
Procedure: Blood Draw — Blood Draw for Troponin Levels - 5ml at baseline and 24 hours later

SUMMARY:
This ancillary study determines whether the Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis (CLOVERS) [ClinicalTrials.gov Identifier: NCT03434028] treatment arms (restrictive fluids strategy vs. liberal fluid strategy) for early sepsis-induced hypotension are associated with differences in cardiac structure and function based on an echocardiogram at 24 hours after randomization. Secondarily, this ancillary study explores possible heterogeneity of treatment effect based on an echocardiogram performed shortly after randomization in CLOVERS.

DETAILED DESCRIPTION:
The Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis: Study of Treatment's Echocardiographic Mechanisms (CLOVERS-STEM) study is an ancillary study to CLOVERS, a parent multi-center, prospective, phase 3 randomized non-blinded interventional trial of fluid treatment strategies in the first 24 hours for patients with sepsis-induced hypotension. The CLOVERS trial attempts to determine the impact of a restrictive fluids strategy (vasopressors first followed by rescue fluids) as compared to a liberal fluid strategy (fluids first followed by rescue vasopressors) on 90-day in-hospital mortality in patients with sepsis-induced hypotension. This ancillary study obtains echocardiograms among CLOVERS-enrolled patients who consent to CLOVERS-STEM at baseline and 24 hours later (secondarily, this study also measures serum troponin levels at baseline and 24 hours) to pursue three aims: 1. Evaluate for differences in left ventricular global longitudinal strain at 24 hours after randomization between treatment arms; 2. Evaluate for differences in right ventricular end diastolic area to left ventricular end diastolic area ratio at 24 hours after randomization between treatment arms; 3. Explore possible heterogeneity of treatment effect based on baseline echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis (CLOVERS) Trial

Exclusion Criteria:

* Lack of Informed Consent for this Ancillary Study
* Allergy to Ultrasound-Enhancing Agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis (CLOVERS) Trial with no allergy to ultrasound-enhancing agents
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Contractility at 24 hours | 24 +/- 6 Hours
  Left Ventricular Global Longitudinal Strain
Right Ventricular Structure at 24 hours | 24 +/- 6 hours
  Right Ventricular End Diastolic Area to Left Ventricular End Diastolic Area Ratio
Day 3 delta SOFA | at 72 hours
  Difference between baseline and day 3 Sequential Organ Failure Assessment (SOFA) scores

SECONDARY OUTCOMES:
Right Ventricular Contractility at 24 hours | 24 +/- 6 hours
  Right Ventricular Longitudinal Strain

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (7):
- United States (7):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health Sciences Center, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected electronically and stored at the Coordinating Center at Intermountain Medical Center. A de-identified version of the analytic data-set will be available for use 3 years after the primary publication. Data can be accessed at that point via the National Heart, Lung and Blood Institute (NHLBI) Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC) data repository.
Time Frame: A de-identified version of the analytic data-set will be available for use 3 years after the primary publication.
Access Criteria: Investigators who complete the appropriate registrations with the Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC) will have access to the de-identified analytic dataset as per BioLINCC policies.
URL: https://biolincc.nhlbi.nih.gov/home/